CLINICAL TRIAL: NCT00044226
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of Two Dosing Regimens of ML-04A in Subjects With Symptomatic Benign Prostatic Hyperplasia
Brief Title: A 20-Week Study of a New Treatment for Men With Benign Prostatic Hyperplasia (BPH).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Milkhaus Laboratory (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ML-BPH-01
Record Dates: First submitted 2002-08-22; First posted 2002-08-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: Prostatic Hyperplasia
Keywords: BPH; Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy; Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia

INTERVENTIONS:
Drug: ML-04A

SUMMARY:
Patients who are currently symptomatic and have been diagnosed with BPH by a physician may qualify for this 20-week study. Patients must not be diabetic, must not have prostate cancer and must not have had any surgery to repair your prostate or treat your BPH. Patients will first undergo a phone screening to confirm their eligibility and interest and to rule out any exclusionary history or medications. Eligible patients will be scheduled to come in to the clinic to sign an Informed Consent Form. Patients will then undergo blood and urine tests, a complete physical examination and history and answer several questionnaires to determine their eligibility. Patients will have a total of at least 7-8 visits over 20 weeks to the clinic during this study.Qualified patients receive free study medication, free medical care (physical examinations, EKG, laboratory tests) for the duration of the study.

DETAILED DESCRIPTION:
Patients must be willing to discontinue their current medications being taken for BPH for specified time periods before they become eligible. These include: Proscar, Saw Palmetto, and any "alpha-blocker" drugs.

Patients with high blood pressure must be on an acceptable medication that controls this condition.

Medications for other conditions may disqualify a patient from eligibility.Patients who are diabetic are not eligible for this study.

All patients will, at some time during the study, receive placebo (inactive substance). The study medication is given twice a day in liquid form under the tongue. There is a 33% chance that you would receive placebo for the duration of the study. Neither you nor your doctor will know which treatment you are receiving.

ELIGIBILITY:
* Have an enlarged prostate by DRE (digital rectal examination);
* Have a diagnosis of BPH;
* Have documented symptoms (frequency; urgency; nighttime urination; reduced flow);
* Have a documented urinary flow rate as required

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2002-04; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Charles White, MD, Mobile, Alabama
  - Douglas Young, MD, Fair Oaks, California
  - Rodney Anderson, MD, Stanford, California
  - Eugene Dula, MD, Van Nuys, California
  - Joel Kaufman, MD, Aurora, Colorado
  - Donald Bergner, MD, Clearwater, Florida
  - Ira Klimberg, MD, Ocala, Florida
  - Gary Friedlander, MD, Rockville, Maryland
  - Sheldon Freedman, MD, Las Vegas, Nevada
  - Edward Loizides, MD, Bay Shore, New York
  - Richard Landau, MD, Sellersville, Pennsylvania
  - H. Pat Hezmall, MD, Fort Worth, Texas
  - Michael Godschalk, MD, Richmond, Virginia
  - Roger Fincher, MD, Spokane, Washington